CLINICAL TRIAL: NCT04876989
Title: The Comparison of Sympathetic Blockade of Stellate Ganglion Block and Thoracic Paravertebral Block in Patients With Chronic Upper Extremity Neuropathic Pain: a Prospective Randomized and Comparative Clinical Trial
Brief Title: The Comparison of Sympathetic Blockade of Stellate Ganglion Block and Thoracic Paravertebral Block
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University (Other)
Collaborators: SMG-SNU Boramae Medical Center (Other)
Responsible Party: Principal Investigator, Jeeyoun Moon, Associate Professor, Seoul National University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2102-183-120
Record Dates: First submitted 2021-05-03; First posted 2021-05-07 (Actual); Last update posted 2023-10-17 (Actual); Status verified 2023-10

CONDITIONS: Complex Regional Pain Syndromes; Postherpetic Neuralgia; Phantom Limb Pain; Chronic Post Surgical Pain; Post-Traumatic Neuralgia; Neuropathic Pain
MeSH Terms: conditions — Complex Regional Pain Syndromes; Neuralgia, Postherpetic; Phantom Limb; Pain, Postoperative; Neuralgia

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- US-SGB (Active Comparator): 5 ml of 1% mepivacaine is injected for stellate ganglion block using the Ultrasound(US)-guided lateral approach at the sixth cervical vertebral level.
  Interventions: Procedure: US-SGB
- US-TPVB (Active Comparator): 10 ml of 1% mepivacaine is injected for thoracic paravertebral block using the Ultrasound(US)-guided sagittal approach at the second thoracic paravertebral space.
  Interventions: Procedure: US-TPVB

INTERVENTIONS:
Procedure: US-SGB — Well trained pain physician performs all the ultrasound(US)-guided stellate ganglion block(SGB)s, who is not involved in evaluating study variables. Electrocardiography, noninvasive blood pressure, heart rate, and peripheral oxygen saturation were monitored for all patients before, while, and after conducting procedure. For US-guided SGB, patients are supine positioned, and skin preparation on injection site is done with chlorohexidine. Procedure is conducted under ultrasound guidance at C6 level. 5 ml of 1% mepivacaine is injected for the US-SGB group.
  Arms: US-SGB
Procedure: US-TPVB — Well trained pain physician performs all the ultrasound(US)-guided thoracic paravertebral block(SGB)s, who is not involved in evaluating study variables. Electrocardiography, noninvasive blood pressure, heart rate, and peripheral oxygen saturation were monitored for all patients before, while, and after conducting procedure. For US-guided TPVB, patients are prone positioned, and skin preparation on injection site is done with chlorohexidine. Procedure is conducted under ultrasound guidance at T2 paravertebral space. 10 ml of 1% mepivacaine is injected for the US-TPVB group.
  Arms: US-TPVB

SUMMARY:
The purpose of this study is to investigate the effect of ultrasound-guided thoracic paravertebral block (TPVB) when performing sympathetic block for upper limb pain control.

DETAILED DESCRIPTION:
Well-trained pain physicians performs all US-guided stellate ganglion block(SGB)s or US-guided thoracic paravertebrl block(TPVB)s, who is not involved in evaluating study variables. Electrocardiography, noninvasive blood pressure, heart rate, and peripheral oxygen saturation were monitored for all patients before, while, and after conducting procedure.

For US-guided SGB, patients are supine positioned, and skin preparation on injection site is done with chlorohexidine. Procedure is conducted under ultrasound guidance at C6 level. 5 ml of 1% mepivacaine is injected for the SGB group. Syringes are prepared by one nurse who do not involved in other steps of this study.

For US-guided TPVB, patients are prone positioned, and skin preparation on injection site is done with chlorohexidine. Procedure is conducted under ultrasound guidance at T2 paravertebral space. 10 ml of 1% mepivacaine is injected for the TPVB group. Syringes are prepared by one nurse who do not involved in other steps of this study.

Temperature measurement is conducted 2 times (before US-guided SGB or TPVB and after 20 minutes) at both hands by one person who's not involved in other measuring in the study.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of complex regional pain syndrome
* Clinical diagnosis of postherpetic neuralgia
* Clinical diagnosis of phantom limb pain
* Clinical diagnosis of chronic post-surgical pain
* Clinical diagnosis of post-traumatic pain syndrome
* Upper extremity pain lasting more than 3 months

Patients with a new or known diagnosis of chronic neuropathic pain lasting more than 3 months in the upper extremity

Exclusion Criteria:

* Refusal of a patient
* Any vascular disease in the upper extremities
* Previous history of thoracic sympathetic or stellate ganglion neurolysis (e.g. -thermocoagulation, radiofrequency neuromodulation, and/or chemical neurolysis)
* Coagulopathy
* Systemic infection or local infection at the needle injection site
* Major deformation at the level of the neck (radiotherapy, surgery, etc.)
* Known allergy to local anesthetics of amide type
* Inability to understand a numeric rating pain scale (cognitive dysfunction)
* Patients whose palm temperature on the ipsilateral side is ≥ 36.5℃ in the thermography before the procedure

Ages: 19 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2021-07-21 (Actual); Primary Completion 2022-12-19 (Actual); Study Completion 2023-01-16 (Actual)

PRIMARY OUTCOMES:
Proportion of patients reaching > 1.5°C rise of temperature in the ipsilateral hand compared to the contralateral hand | 20 minutes after US-guided thoracic paravertebral block or US-guided stellate ganglion block
  Temperature is measured with a laser thermometer on the palmar aspect of 3 cm below from the middle finger.

SECONDARY OUTCOMES:
Difference of temperature change (°C) between ipsilateral hand and contralateral hand | 20 minutes after US-guided thoracic paravertebral block or US-guided stellate ganglion block
  Temperature is measured with a laser thermometer on the palmar aspect of 3 cm below from the middle finger.
Severity of pain | Time before block and 20 minutes and 1 week and 4weeks after US-guided thoracic paravertebral block or US-guided stellate ganglion block
  The severity of the pain will be evaluated before the block and 20 minutes, 1 week and 4 weeks after the block using an 11-pointed NRS (numerical rating scale) pain score.
Patient global impression change (PGIC) | Time 20 minutes and 1 week and 4 weeks after US-guided thoracic paravertebral block or US-guided stellate ganglion block
  The PGIC will be evaluated 20 minutes, 1 week and 4 weeks after the block using a 5-point Likert scale.
Comparison of Korean version CISS(Cold Intolerance Symptom Severity) Questionnaire | Time before block and 4 weeks after US-guided thoracic paravertebral block or US-guided stellate ganglion block
  Check the CISS before the procedure and 4 weeks after the procedure.
Blood flow velocity measurement in upper extremity vessel(ipsilateral brachial artery) using ultrasound | Time before block and 20minutes after US-guided thoracic paravertebral block or US-guided stellate ganglion block
  The blood flow velocity in the ipsilateral brachial artery will be measured before the block and 20 minutes after the block using a Doppler mode ultrasound device.

CONTACTS AND LOCATIONS:
Overall Officials: Youn Moon Jee, MD, PhD, Study Director — Seoul National University Hospital; Jeongsoo Kim, MD, Principal Investigator — SMG-SNU Boramae Medical Center
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No